CLINICAL TRIAL: NCT00783471
Title: Docetaxel Combined With Pulsatile Erlotinib (Tarceva®) In Patients With Metastatic Non Small Cell Lung Cancer (NSCLC) (DOPERLO)
Brief Title: Docetaxel Intermittent-Erlotinib (Tarceva®) In Metastatic Non Small Cell Lung Cancer (NSCLC)
Acronym: DOPERLO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The low accrual rate of the study (30% of the expected accrual rate)/Low efficacy in both treatment arms.
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: G. Fountzilas/President, Hellenic Cooperative Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE 2D/07
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Erlotinib followed by Docetaxel
  Interventions: Drug: Erlotinib, Docetaxel
- 2 (Experimental): Docetaxel followed by Erlotinib
  Interventions: Drug: Docetaxel, Erlotinib

INTERVENTIONS:
Drug: Erlotinib, Docetaxel — Drug: Erlotinib 150 mg po daily, days 1-12 Drug: Docetaxel 75 mg/m2 IV over 30 min on day 15 Treatment will be repeated every 21 days
  Arms: 1
Drug: Docetaxel, Erlotinib — Drug: Docetaxel 75 mg/m2 IV over 30 min on day 1 Drug: Erlotinib 150 mg po daily, days 4-15 Treatment will be repeated every 21 days
  Arms: 2

SUMMARY:
To determine the more effective dosing sequence of intermittent erlotinib and docetaxel for treating patients with the diagnosis of advanced Non-Small-Lung-Cancer

DETAILED DESCRIPTION:
The combination of chemotherapy [such as docetaxel] with continuous administration of targeted drugs which block the molecular machinery of cancer cell growth [such as erlotinib] have failed to improve their efficacy over only-chemotherapy in patients with metastatic lung cancer of the non-small cell histology type. It is not yet known whether administering targeted drugs intermittently could result in improved efficacy of the combinations. This is a multicenter randomized Phase II trial aiming to determine the more active dosing sequence between intermittent erlotinib and docetaxel for treating patients with advanced Non-Small-Lung-Cancer.Patients will be randomly assigned to one of two treatment arms: they will receive a 12-days course of erlotinib either before docetaxel [arm A] or after docetaxel administration [arm B].Treatment will be repeated every 21 days.Patients will be evaluated every 2 cycles (~6 weeks) for response using RECIST criteria. Those patients achieving stable disease or better will continue therapy up to a total 8 cycles. Those patients experiencing progressive disease will be taken off study. Biopsy material will be assessed for biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 to 75 years inclusive, with histologically confirmed metastatic NSCLC will be enrolled.
2. Patients must have not been previously treated with anticancer drugs for advanced disease.
3. ECOG performance status of 0 - 1.
4. Life expectancy of at least 12 weeks.
5. Patients must be able to take oral medication.
6. At least 4 weeks since any prior major surgery or extended-field radiotherapy. Patients who, in the opinion of the investigator, have fully recovered from limited surgery or have undergone limited-field radiotherapy within 2 weeks may also be considered eligible for the study
7. Granulocyte count > 1,500/mm3 and platelet count > 100,000/mm3. Haemoglobin ³ 9.0g/dl.
8. SGOT (AST) and SGPT (ALT) < 2,5 x ULN in the absence of liver metastases or up to 5 x ULN in case of liver metastases
9. Alkaline phosphatase (ALP) < 2,5 x ULN. If alkaline phosphatase is > 2.5 x ULN, SGOT (AST) and SGPT (ALT) must be < 1.5 x ULN. If alkaline phosphatase is ³ 2.5 x ULN in the presence of liver metastases, SGOT and SGPT must be < 5 x ULN
10. Serum creatinine <= 1.5 ULN or creatinine clearance > 60 ml/min.
11. Normal serum calcium.
12. For all females of childbearing potential a negative pregnancy test must be obtained within 48 hours before starting Tarceva/placebo treatment.
13. Patients with reproductive potential must use effective contraception.
14. Able to comply with study and follow-up procedures.
15. Written (signed) Informed Consent to participate in the study.
16. Written (signed) Informed Consent for use of tumour samples.
17. Presence of measurable or evaluable disease (lesions that are present but do not fulfil the criteria for measurable disease).
18. Formalin-fixed, paraffin-embedded tumour tissue samples representative of the tumour will be provided to sponsor within 3 weeks of the patient starting chemotherapy

Exclusion Criteria:

1. Prior exposure to agents directed at the HER axis (e.g. gefitinib, cetuximab, trastuzumab).
2. Prior chemotherapy or therapy with systemic anti-neoplastic therapy (e.g., monoclonal antibody therapy) for advanced disease. Prior surgery and/or localised irradiation is permitted.
3. Patients who have undergone complete tumour resection after responding to platinum based chemotherapy.
4. Any unstable systemic disease (including active infections, significant cardiovascular disease, [including myocardial infarction within the previous year], any significant hepatic, renal or metabolic disease) metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of study medication(s) or that might affect the interpretation of the results or render the patient at high risk from treatment complications.
5. Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
6. Patients are excluded if they have symptomatic brain metastasis or spinal cord compression that has not yet been definitively treated with surgery and/or radiation; patients with CNS metastases with evidence of stable disease (clinically stable imaging) and stable neurologic function are allowed to enter the study.
7. Patients who are at risk (in the investigator's opinion) of transmitting human immunodeficiency virus (HIV) through blood or other body fluids are excluded.
8. Any inflammatory changes of the surface of the eye.
9. Patients who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
10. Nursing and/or pregnant women.
11. Hypersensitivity to erlotinib (Tarceva) or to docetaxel or to any of the excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Assessment every 6 weeks

SECONDARY OUTCOMES:
To compare the Overall Survival (OS),the Objective Response Rate (ORR) and duration of response | Assessment every 6 weeks while on treatment and every 3 months post completion of 8 cycles of treatment until progression
Identify predictive signaling molecules of the EGFR pathway | Assessment every 6 weeks while on treatment and every 3 months post completion of 8 cycles of treatment until progression

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Briasoulis, MD, Principal Investigator — University of Ioannina Hospital, Medical School
Locations (13):
- Greece (13):
  - Sotiria Hospital, Athens
  - "Alexandra" Hospital, Athens
  - "Attikon" University Hospital, 2nd Dept. of Internal Medicine, Propaedeutic, Oncology Section, Athens
  - Agii Anargiri Cancer Hospital, 3rd Dept. of Medical Oncology, Athens
  - Hygeia Hospital, Athens
  - University General Hospital of Ioannina, Medical Oncology Dept, Ioannina
  - Larissa University Hospital, Larissa
  - Metropolitan Hospital, Second Dept of Medical Oncology, Piraeus
  - Metropolitan Hospital, 1st Dept. of Medical Oncology, Pireaus
  - Patras University Hospital, Dept. of Internal Medicine, Oncology Section, Rio, Patras
  - Theagenio Cancer Hospital, 2nd Dept of Medical Oncology, Thessaloniki
  - Theagenio Cancer Hospital, 3rd Dept. of Medical Oncology, Thessaloniki
  - "Papageorgiou" Hospital, Thessaloniki